CLINICAL TRIAL: NCT00336102
Title: Thyroid Function & Breast Cancer: A Pilot Study to Estimate the Prevalence of Thyroid Dysfunction in Women Diagnosed With Breast Cancer and the Magnitude of Change in Thyroid Function Post-Chemotherapy
Brief Title: Thyroid Dysfunction in Women With Newly Diagnosed Breast Cancer Compared to Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: SCUSF 0502; SCUSF-0502 (Other: SunCoast CCOP Research Base); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer; Fatigue; Hypothyroidism
Keywords: fatigue; hypothyroidism; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Hypothyroidism | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Markers of thyroid function including thyroid stimulating hormone (TSH), Free thyroxine (free T4) and Thyroid peroxidase antibody (TPO Ab). These will be performed at baseline, in 12 months and again 24 months after enrollment. All thyroid function marker assays will be performed by LabCorp.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 Breast Cancer Patient Cases: Patients between the ages of 25 and 75, diagnosed with primary, operable, stage I-III B breast cancer with planned chemotherapy regimen Adriamycin / Cytoxan (AC) plus a taxane are trial candidates.
  Will have physiologic testing at baseline to assess thyroid function and fatigue assessment and management inventory. Will follow-up on management of therapy complications for thyroid disorder if one identified or until off study.
  Interventions: Other: physiologic testing; Procedure: fatigue assessment and management; Procedure: management of therapy complications
- Group 2 Healthy Controls: Controls will be women from the same general demographic area as Group 1 Cases, have no prior history of cancer and be within 5 years of the Group 1 case's age (+/- 5 years).
  Will have physiologic testing at baseline to assess thyroid function and fatigue assessment and management inventory. Will follow-up on management of therapy complications for thyroid disorder if one identified or until off study.
  Interventions: Other: physiologic testing; Procedure: fatigue assessment and management; Procedure: management of therapy complications

INTERVENTIONS:
Other: physiologic testing — Markers of thyroid function including thyroid stimulating hormone (TSH), Free thyroxine (free T4) and Thyroid peroxidase antibody (TPO Ab). These will be performed at baseline, in 12 months and again 24 months after enrollment. All thyroid function marker assays will be performed by LabCorp.
  Other Names: thyroid function tests
Procedure: fatigue assessment and management — Fatigue Symptoms Inventory (FSI) survey
  Other Names: FSI; Fatigue Symptoms Inventory
Procedure: management of therapy complications — If baseline testing results suggest hyperthyroidism or hypothyroidism, the enrolling center will give test results to participants for follow-up with their primary healthcare provider. Participants with hypothyroidism, who are not started on thyroid hormone, will continue on study, given the TSH level is below 10. Those with hypothyroidism who have treatment initiated will not continue on study. Participants who develop hypothyroidism during the study will not continue on-study if replacement therapy is initiated or if the TSH level is 10 or higher. Work up the next control nominated by the patient or contact the patient for the name of another control

SUMMARY:
RATIONALE: Learning about thyroid dysfunction in patients with breast cancer may help plan treatment and may help patients live more comfortably.

PURPOSE: This clinical trial is studying how often thyroid dysfunction happens in women with newly diagnosed stage I, stage II, or stage III breast cancer who are planning to undergo chemotherapy compared to how often it happens in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the proportion of hypothyroidism in women with newly diagnosed stage I-IIIB breast cancer (prior to chemotherapy) vs in cancer-free, age-matched healthy volunteers.
* Compare the magnitude of change in thyroid function in these patients from baseline to 24 months vs in cancer-free, age-matched healthy volunteers.

Secondary

* Correlate variation in thyroid function with fatigue symptom scores.
* Correlate variation in thyroid function with anthropometric measurements.

OUTLINE: This is a pilot, multicenter study.

Patients and age-matched healthy volunteers undergo blood collection at baseline and at 12 and 24 months after enrollment. They also undergo anthropometric measurements and complete the Fatigue Symptom Inventory at baseline and at 12 and 24 months after enrollment.

PROJECTED ACCRUAL: A total of 270 patients and 280 healthy volunteers will be accrued for this study.

ELIGIBILITY:
CASE SELECTION:

* CASE INCLUSION CRITERIA:
* Women between the ages of 25 and 75
* Diagnosed with primary and operable Stage I - IIIB breast cancer
* Scheduled to receive neoadjuvant or adjuvant Adriamycin and Cytoxan (AC) plus a taxane (taxane may be given with AC or follow AC)
* No chemotherapy prior to baseline sample collection
* No prior history of other cancers (except non-melanoma skin cancer)
* Preoperative radiation therapy is permitted
* No diagnosis of hypothyroidism or hyperthyroidism.
* CASE EXCLUSION CRITERIA:
* Stage IV breast cancer
* Scheduled to receive neoadjuvant hormonal therapy (patients who will receive adjuvant hormonal therapy may participate)
* Received adjuvant hormonal therapy or chemotherapy prior to sample collection
* On chemotherapeutic regimen other than Adriamycin and Cytoxan plus a taxane.
* Patients receiving monoclonal antibodies or other biologic therapy may not participate
* Patients scheduled to receive Herceptin may not participate
* Diagnosed with hyperthyroidism or hypothyroidism. (Women being treated for hypothyroidism are not eligible)
* Women with a baseline TSH of 10 or higher will not continue on study
* Women who are pregnant or lactating are not eligible. (Women of childbearing potential who are planning to become pregnant within the next 24 months should not enroll in this study)

CONTROL SELECTION:

* CONTROL INCLUSION CRITERIA:
* Cannot be a blood relative of the case. They can be friends, neighbors, women from social activities, local business, doctors' offices, etc.
* Must live near or in the town of the case
* Women between the ages of 20 and 80 (age-matched to cases +/- 5 years)
* No prior history of cancer (except non-melanoma skin cancer)
* Women ages 40 and older should have had a mammogram within 2 years of study entry, showing no evidence of breast cancer.
* The friend control may bring their mammogram report or send a release and have records faxed to the enrolling center.
* Women under the age of 40 should have had a clinical breast examination within 2 years of study entry, showing no need for diagnostic mammography. If a mammogram was required, it should show no evidence of breast cancer.
* The friend control may bring their mammogram / breast exam report or send a release and have records faxed to the enrolling center.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a pilot study with a planned accrual of 270 patients (cases) and 280 healthy volunteers (controls). Patients between the ages of 25 and 75, diagnosed with primary, operable, stage I-III B breast cancer with planned chemotherapy regimen Adriamycin / Cytoxan (AC) plus a taxane are trial candidates. Participants will be asked to nominate 2 women to serve as their healthy control. In the event the first woman is not eligible or decides not to participate, the second woman will be evaluated. Controls will be women from the same general demographic area, have no prior history of cancer and be within 5 years of the patient's age (+/- 5 years).
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2006-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Compare proportion of hypothyroidism in women with newly diagnosed stage I-IIIB breast cancer prior to chemotherapy vs in age-matched healthy volunteers | 2 years
Compare change in thyroid function from baseline to 24 months after enrollment | 2 years

SECONDARY OUTCOMES:
Correlate variation in thyroid function with fatigue symptom scores and anthropometric measurements at baseline and 24 months after enrollment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nagi B. Kumar, PhD RD FADA, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (41):
- United States (41):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Cancer Centers of Central Florida, PA, Leesburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Medical College of Georgia Cancer Center, Augusta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - William Beaumont Hospital - Troy Campus, Troy, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - MBCCOP - Our Lady of Mercy Comprehensive Cancer Center, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Rutherford Internal Medicine Associates, PA, Forest City, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center - Wilson, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - AnMed Cancer Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Scott and White Hospital, Temple, Texas
  - Scott and White Cancer Institute, Temple, Texas